CLINICAL TRIAL: NCT06799325
Title: The Effect of Acceptance and Commitment Therapy-based Stress Management Program on Psychological Flexibility and Caregiver Burden in Caregivers of Schizophrenia Patients
Brief Title: The Effect of Acceptance and Commitment Therapy Intervention on Caregiver Burden in Caregivers of Schizophrenia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, ZARİF GAYE ARSLAN, research assistant, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CU-SBF-ZGA-01
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-03

CONDITIONS: Care Burden; Schizophrenia; Caregiver Mental Health
Keywords: schizophrenia; care burden; acceptance and commitment therapy; stress management; psychological flexibility
MeSH Terms: conditions — Caregiver Burden; Schizophrenia

STUDY DESIGN:
Intervention Model Description: One intervention group and a control group The Acceptance and Commitment Therapy Based Stress Management Program consisting of 6 sessions, 1 session per week and each session lasting 45 minutes, will be applied to the intervention group. At the end of the application (after 6 weeks), the Psychological Flexibility Scale and the Caregiver Burden Scale will be applied to the intervention group. After 6 weeks, in the 1st month, 2nd month and 3rd month, the Psychological Flexibility Scale and the Caregiver Burden Scale will be applied to the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The Stress Management Program Based on Acceptance and Commitment Therapy will be applied to the intervention group, consisting of 6 sessions, 1 session per week, and each session lasting 45 minutes.
  After the program, scales will be applied in the 1st month, 2nd month and 3rd month.
  Interventions: Behavioral: acceptance and commitment therapy based stress management program
- control group (No Intervention): only scales will be applied and no intervention will be made. Following the application of the first scale, scales will be applied at 1 month, 2 months and 3 months.

INTERVENTIONS:
Behavioral: acceptance and commitment therapy based stress management program — The Stress Management Program Based on Acceptance and Commitment Therapy will be applied to the intervention group, consisting of 6 sessions, 1 session per week, and each session lasting 45 minutes.
  Arms: Intervention group

SUMMARY:
The aim of this study was to learn the effects of Acceptance and Commitment Therapy based stress management program on psychological flexibility and caregiver burden in caregivers of schizophrenia patients. This study is a randomized controlled trial. The main questions it aims to answer are:

* Does an acceptance and commitment therapy-based stress management program increase psychological flexibility in caregivers of patients with schizophrenia?
* Does an acceptance and commitment therapy-based stress management program reduce caregiver burden in caregivers of schizophrenia patients?
* What is the relationship between the level of psychological flexibility and care burden? Researchers will compare the intervention with a control group (no intervention) to see if an acceptance and commitment therapy-based stress management program increases psychological resilience and reduces caregiver burden in people with schizophrenia.

Participants will participate in the Acceptance and Commitment Therapy Based Stress Management Program, consisting of 6 sessions, one session per week, each session lasting 45 minutes.

The intervention group will visit the clinic at the end of the application (after 6 weeks), at 1 month, 2 months and 3 months to be administered the Psychological Flexibility Scale and the Caregiver Burden Scale.

They will do the homework given in the therapy program.

DETAILED DESCRIPTION:
Approximately 25-50% of schizophrenia patients worldwide, and 70% of schizophrenia patients in Asia, live with their families. Schizophrenia-related symptoms affect the individual as well as their family and caregivers. The severity of disease symptoms and the decrease in productivity of patients increase the care burden of family members and affect their physical and psychological health. Caring for patients with schizophrenia is a difficult, sensitive, and time-consuming responsibility. Caregiving creates social, emotional, behavioral, and financial problems for caregivers and causes various limitations in their personal lives. Caregivers of patients with schizophrenia are at serious risk of caregiver burden and psychiatric morbidity.Caregivers of schizophrenia patients experience high levels of caregiver burden and stress. It has been reported that family interventions reduce the relapse rate and hospitalization time in schizophrenia, and increase the duration of remission. Therefore, implementation of interventions that reduce the caregiver burden is very important to provide the best care for the patient, while also preventing mental illnesses that may develop in family caregivers. Developing stress coping methods and psychological flexibility of caregivers of schizophrenia patients with an acceptance and commitment therapy-based stress management program may be effective in reducing the caregiver burden. It is thought that with the implementation of this program, caregivers will develop more effective coping behaviors against stress, and in parallel, the risk of caregiver burden, stress, and mental illness will decrease.

This research is a randomized controlled trial to determine the effects of an individual Acceptance and Commitment therapy-based stress management program on psychological flexibility and caregiver burden in caregivers of schizophrenia patients.

Research Hypothesis/Hypotheses H1. At the end of the application of the acceptance and commitment therapy based stress management program, there is a difference between the intervention and control group psychological flexibility scores.

H2. At the end of the application of the acceptance and commitment therapy based stress management program, there is a difference between the intervention and control group care burden scores.

H3. At the end of the application of the acceptance and commitment therapy based stress management program, there is a difference between the intervention and control group care burden scores in the first, second and third months.

H4. At the end of the application of the acceptance and commitment therapy based stress management program, there is a difference between the intervention and control group psychological flexibility scores in the first, second and third months.

The Universe and Sample of the Study The universe of this study will consist of the caregivers of patients diagnosed with schizophrenia who were hospitalized in Sivas Hospital and Sivas Cumhuriyet University Application and Research Hospital psychiatry clinic between March 22, 2024 and March 01, 2025. The number of patients to be included in the study sample was determined by performing power analysis with the G-Power 3.1.9.4 sample volume calculation program. Accordingly, when the standard deviation was one, the effect size was 0.76, the significance level was 0.05 and (1-β)=0.80, the power of the study was calculated as 0.80678. The sample size will consist of the caregivers of 60 patients. 30 of the caregivers will form the intervention group (n1) and 30 will form the control group (n2).

Measurement Tools Used in the Study

1. Personal Information Form:
2. Psychological Flexibility Scale:
3. Caregiver Burden Scale:
4. DISCERN (Quality Criteria for Consumer Health Information) Scale: It was to be used in the evaluation of the content and quality of educational materials. The DISCERN measurement tool, which consists of three sections, includes 16 questions that question the content of the material.

Obtaining Expert Opinions A total of 5 expert opinions were obtained regarding the acceptance and commitment therapy-based stress management guide, including 3 faculty members specialized in psychiatric nursing, 1 faculty member specialized in public health and 1 faculty member specialized in clinical psychology. The experts were asked to evaluate the prepared guide in accordance with the Written Materials Appropriateness Evaluation Form and the DISCERN Scale. The expert opinions evaluated with the DISCERN Scale were analyzed. The intervention program was finalized in line with the opinions. The preliminary application of the research was carried out and changes were made regarding the aspects that needed to be adjusted.

Research Process The research will be conducted in the psychiatry clinics of Sivas Hospital and Sivas Cumhuriyet University Hospital. Caregivers of schizophrenia patients receiving inpatient treatment will be interviewed in the interview room of the psychiatry clinic between the research dates. Consent forms will be obtained from those who want to participate in the study and the study will be conducted on caregivers who meet the participation criteria. Individuals who agree to participate in the study will be assigned to the intervention and control groups through randomization. The first interview will be conducted with the intervention and control groups and the Psychological Flexibility Scale, Caregiver Burden Scale and Personal Information Form will be filled out.

The intervention group will be informed about the program and its goals. The Acceptance and Commitment Therapy Based Stress Management Program consisting of 6 sessions, 1 session per week and each session lasting 45 minutes, will be applied to the intervention group.

The purpose of the research will be explained to the control group and it will be stated that the scales will be applied at certain intervals within the scope of this research and measurements will be made simultaneously with the intervention group.

No program will be applied to the control group during the application and follow-up periods.

At the end of the application (after 6 weeks), the psychological flexibility scale and the caregiver burden scale will be applied to the intervention and control groups in the 1st month, 2nd month and 3rd month.

Data Analysis The data obtained from our study will be loaded into the Statistical Package for the Social Sciences program (Ver: 22.0) and when the parametric test assumptions are met (Kolmogorov Smirnov), Variance Analysis, Bonferroni test, significance test of the difference between two means will be used in repeated measurements, and when the parametric test assumptions are not met, Friedman test, Wilcoxon test, Mann Whitney U test and Chi-square test will be used and the error level will be taken as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65,
* A primary caregiver of a patient diagnosed with schizophrenia according to -
* Diagnostic and statistical manual of mental disorders- V for more than 1 year,
* A person who has lived in the same house with the patient for at least 6 months and is primarily responsible for the patient's care,
* A person who has at least a secondary school degree,
* A person who can communicate verbally

Exclusion Criteria:

* Individuals with mental illness,
* Individuals who do not live in the same house as the patient,
* Individuals with perception and communication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Caregiver Burden Scale | 6 weeks after registration, In the 1st month, in the 2nd month, in the 3rd month
  The scale consists of a total of 22 statements to determine the level of impact on the lives of caregivers. The scale, which can be completed in a question-answer format by the caregiver at home or with the researcher, has a Likert-type assessment ranging from 0 to 4 as never, rarely, sometimes, often, or almost always. The minimum score from the scale is 0, while the maximum score is 88. The items in the scale are mostly social and emotional, and a high scale score indicates high distress. The reliability study of the scale, which has been used by different researchers in Turkey, was translated by İnci and colleagues in 2006. The Cronbach alpha value indicating the reliability coefficient was found to be 0.95 for the Caregiver Burden Scale, indicating a high level of reliability.

SECONDARY OUTCOMES:
Psychological Flexibility Scale | 6 weeks after registration, In the 1st month, in the 2nd month, in the 3rd month
  Validity study and Turkish adaptation of the scale were conducted and Cronbach's Alpha internal consistency reliability coefficient was found to be .79. The scale consists of 28 items and 5 sub-dimensions. It is a 7-point Likert-type scale. Items 2, 3, 5, 6, 8, 18, 20, 22, 23, 24 and 25 are scored reversely. The lowest score that can be obtained from the scale is 28, and the highest score is 196. In the evaluation of the scale items, high scores obtained from each sub-scale indicate that individuals are psychologically flexible.

CONTACTS AND LOCATIONS:
Overall Officials: havva tel, Professor, Study Director — havatel@cumhuriyet.edu.tr
Locations (1):
- Sivas Cumhuriyet University Faculty of Health Sciences Nursing Department, Sivas, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No